CLINICAL TRIAL: NCT04947904
Title: Impact on Fluid Balance of an Optimised Restrictive Strategy Targeting Non-Resuscitative Fluids in Intensive Care Patients Hospitalised for Septic Shock: an Open-label, Multi-Centre, Randomised, Controlled Pilot Study.
Brief Title: OPTImized Restrictive Strategy Targeting Non-Resuscitative FLUIDs in Septic Shock: Pilot Study.
Acronym: OPTIFLUID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: University Hospital, Montpellier (Other); Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NIMAO/2019/SB-01; 2020-A01952-37 (Other: ANSM)
Record Dates: First submitted 2021-06-14; First posted 2021-07-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Septic Shock; Electrolyte and Fluid Balance Conditions
Keywords: Shock, Septic.; Fluid Balance
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimised Restrictive Strategy (Experimental): The volume of non-resuscitative fluids infused to the patient will be reduced by the doctor in charge of the patient for the first 7 days of the patient's stay in ICU according to a special protocol.
  Interventions: Other: Reduction of the patient's fluid intake during the first 7 days
- Control (No Intervention): Resuscitation fluids, maintenance fluids, nutrition and drugs will be administered as usually performed and following most recent guidelines.

INTERVENTIONS:
Other: Reduction of the patient's fluid intake during the first 7 days — The volume of fluids infused to the patient will be reduced by the doctor in charge of the patient for the first 7 days of the patient's stay in the intensive care unit according to a protocol with instructions to reduce fluid intake as far as possible in terms of maintenance fluids, dilution of medication and artificial nutrition. This protocol will be begun immediately following the patient's inclusion on Day 1 and pursued for 7 days after inclusion (i.e. from Day 1 - to Day 7). The fluid restriction strategy does not involve the administration of any medication (i.e. diuretics). A clinical pharmacist will help the intensive care teams apply the fluid restriction protocol with a daily check. If the restrictive strategy leads to hypovolemia and / or a electrolyte anomaly (sodium, potassium, chloride, etc.), the physician in charge will be authorised to treat these anomalies in conformance with the protocol recommendations.
  Arms: Optimised Restrictive Strategy

SUMMARY:
Intravenous fluids are one of the keystones in the initial management of patients with septic shock, but they inevitably lead to a fluid overload, which is associated with poor outcome.

So far no studies have evaluated the interest of a restrictive strategy for managing fluid intake targeting all non-resuscitative fluids (fluids for maintenance and drug dilution as well as nutrition) and especially the impact of this restrictive strategy on fluid overload.

The hypothesis of this research is that an optimised restrictive strategy targeting all non-resuscitative fluids in patients hospitalised in the intensive care unit for septic shock, will have an impact on fluid balance in these patients.

DETAILED DESCRIPTION:
Sepsis and its most severe form, septic shock, are the cause of nearly 30% of admission in intensive care unit (ICU). The related mortality rate varies from 20 to 60% according to the studied population and the type of the study. With the concomitant and rapid treatment of the source of infection, hemodynamic optimization with fluid infusion (fluid resuscitation) is the cornerstone of management of patients in septic shock. Nevertheless, fluid overload has been shown to be associated with poor outcome. The negative effects of a positive fluid balance on ICU outcomes for septic patients has been well established.

In patients with acute respiratory distress syndrome, a restrictive fluid therapy has been associated with shorter use of mechanical ventilation. In patients with acute renal failure, fluid overload is associated with longer need of renal replacement therapy. In patients with septic shock numerous non-randomised studies reported that a positive fluid balance at Day 3, Day 5 was associated with an increased risk of mortality.

Actually, in patients with septic shock the part of resuscitation fluid is only the third of the total fluid input that can attain 25 liters at day 3. Some studies reported more specifically the role of the different types of fluid in the fluid balance at D3 and D5. In a retrospective single centre study including 14654 ICU patients over 10 years, the authors distinguished resuscitation, replacement and maintenance fluids, blood products, nutrition and fluid creep (to concentrate electrolytes, keep venous access and to infuse continuous medications). They reported that maintenance fluids and fluid creep represent more than 50% of fluid input during the first 5 ICU days with significant sodium and chloride loads. In a retrospective multi-centre study involving 400 patients mechanically ventilated > 24 h in 10 ICUs, the authors reported that maintenance and fluid creep represented more than 50% of the fluids infused during the first 3 ICU days. In this study, fluid balance at Day3 was an independent risk factor for 30-day mortality.

All these findings could lead to hypothesize that a restrictive strategy in fluid input for the maintenance of fluid and creep fluid could be associated with a better outcome without impairing the resuscitation phase.

To our knowledge, to date, no study has focused on a restrictive strategy targeting non-resuscitative fluid input to optimize fluid balance in patients with septic shock. OPTIFLUID will be the first randomised controlled trial with the objective of reducing fluid balance through a fluid restriction targeted at all fluids other than resuscitative fluids.

The only existing interventional studies on targeted restriction were limited to resuscitative intravenous fluids, and they failed showing a benefit.

By optimizing fluid therapy, our approach is likely to improve patient-centred outcomes, but in this pilot study we focus only on the fluid balance and the safety.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from an infection already documented or suspected
* Patient with organ dysfunction defined as an acute change in SOFA score ≥ 2 points
* Patient with refractory hypotension requiring vasopressors to maintain a mean arterial pressure ≥ 65 mm Hg in spite of resuscitation with an adequate volume of intravenous fluids (according to the recommendations of the Surviving Sepsis campaign). The treatment by vasopressor must have been started less than 24 hours before inclusion and randomization.
* Patient with hyperlactatemia (blood lactate > 2 mmol / L). This criterion must be fulfilled at least once for the purpose of the diagnosis within the 24 hours preceding inclusion and randomization.
* Patient or close relative / legal representative / family member / curator / tutor must have given written informed consent and signed the consent form for the patient included in an emergency situation
* Patient must be covered by a health insurance scheme.
* Adult patient (≥18 years) under 85 years old (< 85).

Exclusion Criteria:

* Patient who has had a previous episode of septic shock requiring vasopressor administration or mechanical ventilation or renal replacement therapy during the current ICU stay.
* A patient whose life expectancy is shortened due to his/her initial health condition or a moribund patient whose life expectancy is less than 48 hours or whose decision to limit comprehensive care was made before including the patient.
* Patient who has had a recent cardiac arrest (during current hospital stay)
* Patient requiring emergency renal-replacement therapy (hyperkalemia [potassium > 6.5 mmol/l] refractory to medical treatment and/or metabolic acidosis [pH <7.15 and partial pressure of carbon dioxide (pCO2) <45 mmHg] refractory to medical treatment and/or pulmonary edema in anuric patients who do not respond to diuretic therapy).
* Patient with KDIGO 3 acute kidney injury and likely to require renal-replacement therapy within the next 24 hours, as determined by the patient's clinician in charge
* Patients with end-stage chronic renal failure or patients already undergoing chronic dialysis
* Severely malnourished patient in whom nutritional support is an emergency procedure (body mass index <18 kg / m2)
* Patient participating in or having participated in an interventional study with similar patient outcome in the previous 3 months.
* Patient in an exclusion period determined by another study.
* Patient under legal protection.
* Pregnant patient (positive serum pregnancy test).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Fluid balance at day 5 | Day 5
  Fluid intakes are noted on a daily basis (parenteral, enteral, and oral routes) and all outgoing fluids (diuresis, depletion on renal-replacement therapy, drainage, diarrhoea (if the volume is measurable). The difference between these daily fluid intakes and outgoing fluids is the daily fluid balance. Fluid balance on Day 5 is the sum total of the fluid balances from Days 1 to 5 and is measured in millilitres per kgs of patient's weight at baseline.

SECONDARY OUTCOMES:
Change from baseline in fluid balance at day 7 | Day 1 to 7
  Fluid intakes are noted on a daily basis (parenteral, enteral, and oral routes) and all outgoing fluids (diuresis, depletion on renal-replacement therapy, drainage, diarrhoea (if the volume is measurable). The difference between these daily fluid intakes and outgoing fluids is the daily fluid balance. Fluid balance on Day 5 is the sum total of the fluid balances from Days 1 to 7 and is measured in millilitres per kgs of patient's weight at baseline.
Change from baseline in patient's weight at day 5 | Day 1 to 5
  The patient's weight will be recorded every day in kgs. The difference in the patient's weight between Day 1 and Day 5 will be recorded in kgs.
Change from baseline in patient's weight at day 7 | Day 1 to 7
  The patient's weight will be recorded every day in kgs. The difference in the patient's weight between Day 1 and Day 7 will be recorded in kgs.
Change from baseline in central venous pressure at day 5 | Day 1 to 5
  Central venous pressure will be recorded every day in mmHg
Change from baseline in central venous pressure at day 7 | Day 1 to 7
  Central venous pressure will be recorded every day in mmHg
Vital status at Day 7 | Day 7
  The number of patients still alive on Day 7 will be recorded
Vital status at Day 28 | Day 28
  The number of patients still alive on Day 28 will be recorded
Proportion of patients alive without organ failure at Day 7 | Day 7
  The Sequential Organ Failure Assessment (SOFA) score will be used will be used to record the patient's condition. The score ranges from 0 to 3 points : one point for each of Low blood pressure (SBP ≤ 100 mmHg), High respiratory rate (≥ 22 breaths/min) and Altered mentation (GCS ≤ 14).The presence of 2 or more SOFA points near the onset of infection was associated with a greater risk of death or prolonged intensive care unit stay. These are outcomes that are more common in infected patients who may be septic than those with uncomplicated infection. The number of patients with a SOFA score = 0 will be recorded.
Proportion of patients alive without organ failure at Day 28 | Day 28
  The Sequential Organ Failure Assessment (SOFA) score will be used to record the patient's condition. The score ranges from 0 to 3 points : one point for each of Low blood pressure (SBP ≤ 100 mmHg), High respiratory rate (≥ 22 breaths/min) and Altered mentation (GCS ≤ 14).The presence of 2 or more SOFA points near the onset of infection was associated with a greater risk of death or prolonged intensive care unit stay. These are outcomes that are more common in infected patients who may be septic than those with uncomplicated infection. The number of patients with a SOFA score = 0 will be recorded.
Vasopressors free days | Day 28
  The number of days the patient has survived without the use of vasopressors will be recorded.
Invasive mechanical ventilation free days | Day 28
  The number of days the patient has survived without the use of invasive mechanical ventilation will be recorded.
Renal-Replacement Therapy free days | Day 28
  The number of days the patient has survived without the use of renal-replacement therapy will be recorded.
Intensive Care Unit Length of stay | Day 28
  The total number of days spent in the ICU will be recorded.
Intensive Care Unit Free Days | Day 28
  The number of days spent in hospital outside the intensive care unit will be recorded.
Hospital Length of stay | Day 28
  The total number of days spent in hospital will be recorded.
Frequency of metabolic disorders - moderate hypernatremia | Day 7
  The frequency of moderate hypernatremia will be recorded to evaluate the safety and tolerance of adverse events associated with the optimal restrictive strategy. Moderate hypernatremia = natremia between 146 and 150 mmol/l.
Frequency of metabolic disorders - severe hypernatremia | Day 7
  The frequency of severe hypernatremia will be recorded to evaluate the safety and tolerance of adverse events associated with the optimal restrictive strategy. Severe hypernatremia = natremia over 150 mmol/l.
Frequency of metabolic disorders - hyponatremia | Day 7
  The frequency of hyponatremia will be recorded to evaluate the safety and tolerance of adverse events associated with the optimal restrictive strategy. Hyponatremia = natremia below 130 mmol/l
Frequency of metabolic disorders - hyperkalemia | Day 7
  The frequency of hyperkalemia will be recorded to evaluate the safety and tolerance of adverse events associated with the optimal restrictive strategy (hyperkalemia over 6 mmol/l
Frequency of metabolic disorders - hypoglycemia | Day 7
  The frequency of hypoglycemia < 0.6g/l will be recorded to evaluate the safety and tolerance of adverse events associated with the optimal restrictive strategy.
Insulin cumulative dose at Day 7 | Day 7
  The cumulative dose of insulin administered over 7 days will be recorded.
Frequency of moderate acute kidney injury | Day 7
  The frequency of moderate acute kidney injury defined by the Kidney Disease Improving Global Outcomes (KDIGO) score 2 will be recorded.
Frequency of severe acute kidney injury | Day 7
  The frequency of severe acute kidney injury defined by the Kidney Disease Improving Global Outcomes (KDIGO) score 3 will be recorded.
Cumulative dose of diuretics at day 7 | Day 7
  The cumulative dose of diuretics administered over 7 days will be recorded.
Frequency of Stage 3 pressure sores | Day 7
  The frequency of Stage 3 pressure sores acquired in the resuscitation unit will be recorded.
Daily fluid intake: Resuscitation Fluids | Day 1 to 7
  The daily volume of crystalloids and colloids supplied to the patient will be recorded daily in milliliters per kilograms of patient's weight
Daily fluids intake: Blood Transfusions and Blood Derivatives | Day 1 to 7
  The daily volume of blood transfusions, Blood Derivatives and plasma-derived products supplied to the patient will be recorded daily in milliliters per kilograms of patient's weight
Daily fluids intake: Maintenance Fluids | Day 1 to 7
  The amount of Maintenance fluids (prescribed to provide water and electrolytes when patients are unable to ingest food or fluids) will be recorded daily in milliliters per kilograms of patient's weight
Daily fluids intake: Fluid Creep | Day 1 to 7
  The volume of fluids administered unintentionally as a vehicle for intravenous, oral, or enteral medication will be recorded daily in milliliters per kilograms of patient's weight
Daily fluids intake : Enteral Nutrition | Day 1 to 7
  The amount of fluid in terms of enteral nutrition will be recorded daily in milliliters per kilograms of patient's weight
Daily fluids intake : Parenteral Nutrition | Day 1 to 7
  The amount of fluid in terms of parenteral nutrition will be recorded daily in milliliters per kilograms of patient's weight
Daily fluids intake : Water | Day 1 to 7
  The volume of water in terms of oral intake and the volume administered in the nasogastric tube will be recorded daily in milliliters per kilograms of patient's weight
Daily fluids intake : intravenous fluids to treat hypernatremia | Day 1 to 7
  The amount of fluids given intravenously to treat hypernatremia (intravenous hydration with a 2.5% glucose solution) will be recorded daily in milliliters per kilograms of patient's weight

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Hospitalier d'Alès, Alès
  - CHU de DIJON, Dijon
  - CHU de Montpellier, Montpellier
  - Nimes University Hospital, Nîmes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Boulet N, Quenot JP, Serrand C, Antier N, Garnier S, Buzancais A, Muller L, Roger C, Lefrant JY, Barbar SD. Impact on fluid balance of an optimized restrictive strategy targeting non-resuscitative fluids in intensive care patients with septic shock: a single-blind, multicenter, randomized, controlled, pilot study. Crit Care. 2024 Dec 21;28(1):429. doi: 10.1186/s13054-024-05155-z. PMID 39709493